CLINICAL TRIAL: NCT07342751
Title: The Effect of Listening to Music During Mobilization on Pain and Fear in Children Undergoing Abdominal Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Assoc. Prof, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22102025
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pain; Surgery; Children, Only
Keywords: pain; mobilisation; surgery; children
MeSH Terms: conditions — Pain | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music (Experimental): Children in this group will be played their preferred and favorite music immediately before the mobilization process begins. The music will continue uninterrupted throughout the mobilization process and will end when the child returns to their bed after mobilization.
  Interventions: Other: music
- control (No Intervention): Children in this group will not receive any musical entertainment; instead, mobilization will be carried out in accordance with the clinic's existing routine procedures, with parental support.

INTERVENTIONS:
Other: music — Children in this group will be introduced to music of their choice and preference immediately before the mobilization begins.
  Arms: music

SUMMARY:
This research is designed to improve the mobilization process in children aged 4-6 years undergoing abdominal surgery. The main objective of the study is to determine the effect of music listening on pain and fear levels in children who are standing up for the first time after surgery using a randomized controlled experimental method. This study, to be conducted at the Pediatric Surgery Department of Aksaray Training and Research Hospital, will involve a total of 74 children (37 in the study group and 37 in the control group) between January 2026 and November 2026.

According to the research protocol, children in the study group will listen to music of their own choosing during mobilization, while children in the control group will receive routine parental support from the clinic. During the data collection process, children's pain levels will be recorded using the Wong-Baker Pain Scale, and their fear levels using the Child Fear Scale, along with assessments from the child, parent, and nurse. Vital signs such as heart rate and respiratory rate will also be monitored before and after the procedure. This study aims to facilitate early mobilization in children and provide evidence as an effective non-pharmacological method in nursing care.

DETAILED DESCRIPTION:
This randomized controlled experimental study aims to investigate the impact of music intervention on the pain and fear levels of children during the postoperative mobilization. Mobilization is a critical part of recovery, but it is often delayed in pediatric patients due to factors such as age, anxiety, fear, and pain. The study is designed to provide evidence for nurses on the use of non-pharmacological methods to facilitate early mobilization and improve the quality of surgical care.The research will be conducted at the Aksaray Training and Research Hospital Pediatric Surgery Department between January 2026 and November 2026. The study population consists of 74 children aged 4-6 who have undergone abdominal surgery. Participants will be randomly and equally divided into two groups: a study group (n=37) and a control group (n=37) using a computer-generated randomization program. Inclusion criteria require that the children be undergoing their first postoperative mobilization, have received only a single dose of paracetamol, and have no chronic illnesses or sensory impairments.The methodology involves assessing both groups before and after the mobilization process. Prior to mobilization, the baseline vital signs (heart rate, respiration, etc.) and pain and fear levels of all children will be evaluated by the child, their parents, and a nurse. During the mobilization, the study group will listen to music of their own choice through headphones, while the control group will receive standard clinical care with parental support. Immediately after the child returns to bed, the evaluations and vital sign recordings will be repeated to measure the intervention's effect.To ensure rigorous data collection, the researchers will use the Wong-Baker FACES Pain Rating Scale, the Children's Fear Scale (CFS), and a Vital Signs Tracking Form. Statistical analysis will be performed using SPSS 25.0, utilizing tests such as independent t-tests, Mann-Whitney U, and Chi-square to determine the significance of the results (p < .05). The study anticipates that the music intervention will significantly lower pain and fear scores, supporting the hypothesis that music is an effective supportive tool in pediatric surgical nursing.

ELIGIBILITY:
Inclusion Criteria:

* Being between 4-6 years old
* Having undergone abdominal surgery
* Having undergone surgery under general anesthesia
* Having received a single dose of analgesic (paracetamol) after surgery
* Having undergone initial mobilization after surgery
* Being a volunteer to participate in the study

Exclusion Criteria:

* Having undergone previous surgery
* Having a chronic illness
* A parent having undergone abdominal surgery
* The child having visual, hearing, physical, or intellectual disabilities

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Wong-Baker Scale | 1 day
  The Wong-Baker Scale was developed by Donna Wong and Connie Morain Baker in 1981 and revised in 1983 to assess children's pain levels. It features six facial expressions scored from zero to five. The Wong-Baker Scale includes faces representing increasing pain intensity from zero to five, from left to right.
Fear Scale | 1 day
  Developed by McMurtry et al. in 2011, it is a scale used to determine the anxiety/fear levels of children. The scale uses five picture faces. Fear level is evaluated with numbers between '0' and '4'. The first picture represents a score of '0', meaning 'no fear felt', and the fifth picture represents a score of '4', meaning 'severe fear'. As the score increases, the level of fear also increases (McMurtry et al., 2011; 780-788; Gerçeker et al., 2018:9-13). The translation and reliability study of the Child Fear Scale into Turkish was carried out by Özalp Gerçeker and colleagues in 2017.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christiaens, G. (2003). Independent nursing interventions for pain management. Home health care management &practice, 15(3), 212-214.
- [Background] Cote, C. J., & Wilson, S. (2016). Guidelinesformonitoringandmanagement of pediatricpatientsbefore, during, andaftersedationfordiagnosticandtherapeuticprocedures: update 2016. PediatricDentistry, 38(4), E19-E39.
- [Background] Gerçeker, G. Ö., Ayar, D., Özdemir, Z., & Bektaş, M. (2018). Çocuk anksiyete skalası-durumluluk ve çocuk korku ölçeğinin Türk diline kazandırılması. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 11(1), 9-13
- [Background] Jones RA, Merkle S, Ruvalcaba L, Ashton P, Bailey C, Lopez M. Nurse-Led Mobility Program: Driving a Culture of Early Mobilization in Medical-Surgical Nursing. J Nurs Care Qual. 2020 Jan/Mar;35(1):20-26. doi: 10.1097/NCQ.0000000000000404. PMID 30889084
- [Background] Gıynaş, T., Önel, A. E., Küçük, S., Uğur, S., & Yardımcı, F. An Investigation of Using Non-PharmacologicalMethods in Pain Management in PostoperativePeriod in Children: A SystematicReview. Bilecik Şeyh Edebali Üniversitesi Sağlık Bilimleri Fakültesi Dergisi, 2(3), 172-190.
- [Background] Sayar, S., & Ergin, D. (2019). Ortopedi servisinde yatan çocuk hastalarda ameliyat sonrası ağrı yönetiminde müziğin etkisinin incelenmesi. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 12(1), 67-73.
- [Background] Kwekkeboom KL, Gretarsdottir E. Systematic review of relaxation interventions for pain. J Nurs Scholarsh. 2006;38(3):269-77. doi: 10.1111/j.1547-5069.2006.00113.x. PMID 17044345